CLINICAL TRIAL: NCT01617382
Title: Register With Data From Patients With the Diagnosis of a Peritoneal Surface Malignancy, for Which Cytoreductive Surgery and Hyperthermic Intra-Peritoneal Chemotherapy (HIPEC) is Performed
Brief Title: Register With Patients in Which Hyperthermic Intra-Peritoneal Chemotherapy (HIPEC) Was Performed
Acronym: HIPEC
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S-54350
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Peritoneal Carcinomatosis; Pseudomyxoma Peritonei; Peritoneal Mesothelioma
Keywords: HIPEC; Hyperthermic (heated) chemotherapy after debulking
MeSH Terms: conditions — Peritoneal Neoplasms; Pseudomyxoma Peritonei; Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Registry: Patients with peritoneal carcinomatosis of colorectal origin, patients with pseudomyxoma peritonei (type DPAM or PMCA) and patients with peritoneal mesothelioma who are planned to undergo cytoreductive surgery and HIPEC because of a peritoneal surface malignancy

SUMMARY:
The purpose of this study is to register the follow-up data of patients who, because of a peritoneal surface malignancy, will undergo cytoreductive surgery and HIPEC.

DETAILED DESCRIPTION:
To register the follow-up data of patients who, because of a peritoneal surface malignancy, will undergo cytoreductive surgery and HIPEC. In this surgical intervention, the abdominal cavity is macroscopically cleared of tumor, by removing all visible tumor nodules, and is subsequently rinsed with hyperthermic (heated) chemotherapy, aiming to destroy all residual invisible tumor cells that might have stayed behind after the debulking.

The eventual aim of this procedure is to improve the prognosis/survival of patients with malignancies localized on the peritoneal surface.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peritoneal carcinomatosis of colorectal origin, patients with pseudomyxoma peritonei (type DPAM or PMCA) and patients with peritoneal mesothelioma who are planned to undergo cytoreductive surgery and HIPEC because of a peritoneal surface malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with peritoneal carcinomatosis of colorectal origin, patients with pseudomyxoma peritonei (type DPAM or PMCA) and patients with peritoneal mesothelioma who are planned to undergo cytoreductive surgery and HIPEC because of a peritoneal surface malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2012-05; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To improve the prognosis/survival of patients with malignancies localized on the peritoneal surface. | Follow-up over a time period of at least 5 years

CONTACTS AND LOCATIONS:
Overall Officials: André JL D'Hoore, PhD, Principal Investigator — University Clinics Gasthuisberg Department of Abdominal Surgery
Locations (1):
- University Clinics Gasthuisberg, Leuven, Flemish Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No